CLINICAL TRIAL: NCT01617304
Title: Effects of Food Cooking on Diabetes-2 Risk Factors
Acronym: Age-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: The Ministry of Science, Technology and Innovation, Denmark (Other Government)
Responsible Party: Principal Investigator, AAstrup, Head of Department, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: M201
Record Dates: First submitted 2012-02-22; First posted 2012-06-12 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Obesity; Type 2 Diabetes; Insulin Resistance; Cardiovascular Disease
Keywords: advanced glycation end products; insulin sensitivity; obesity; inflammation; metabolomics; appetite; CVD
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Insulin Resistance; Cardiovascular Diseases; Inflammation | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- low AGE, glucose (Experimental): Food prepared by boiling/steaming and 20 g of glucose 3 times a day in a water solution
  Interventions: Other: Dietary intervention
- low AGE, fructose (Experimental): Food prepared by boiling/steaming and 20 g of fructose 3 times a day in a water solution
  Interventions: Other: Dietary intervention
- high AGE, fructose (Experimental): Food prepared by frying/baking and 20 g of fructose 3 times a day in a water solution
  Interventions: Other: Dietary intervention
- high AGE, glucose (Experimental): Food prepared by frying/baking and 20 g of glucose 3 times a day in a water solution
  Interventions: Other: Dietary intervention

INTERVENTIONS:
Other: Dietary intervention — Food made by different cooking methods (boiling/steaming versus frying) and with glucose or fructose water solution

SUMMARY:
The aim of the project is to investigate the effects of advanced glycation end products (AGEs) formed in food during the cooking process as well as AGEs formed naturally in the human body, on insulin sensitivity and risk factors for type 2 diabetes. The hypothesis is that i) food content of AGEs is lower using boiling and steaming cooking methods and that ii) AGEs formation in the body is lower at low dietary intake of certain sugar forms.

ELIGIBILITY:
Inclusion Criteria:

* women, healthy between 20 and 50 y
* BMI between 25 and 40 kg/m2
* weight circumference over 88 cm

Exclusion Criteria:

* weigh changes within the last 2 months more than +/- 3 kg
* Physical activity more than 8 h per week
* smoking
* medications and supplements
* being vegetarian or vegan
* pregnancy or breast feeding
* postmenopause
* chronic disease
* previous gastric bypass surgery
* blood donation within the last 3 months
* Involvement in other clinical trials
* allergic to paraaminobenzoic acid

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
change in HOMA from baseline to 4 weeks | 0 and 4 weeks
  insulin sensitivity
change in OGTT from baseline to 4 weeks | 0 and 4 weeks at 0 and 120 min
  insulin sensitivity
change in appetite hormones (leptin, adiponectin, GLP-1, glukagon, ghrelin) from baseline to 4 weeks | 0 and 4 weeks
change in plasma and urin AGEs from baseline to 4 weeks | 0 and 4 weeks
change in immune response (CRP, C-peptide, IL-1B, IL-6, VCAM, ICAM, MIF, TNF-a, buffycoat) from baseline to 4 weeks | 0 and 4 weeks
change in metabolomics dats from baseline to 4 weeks | 0 and 4 weeks
change in AGE levels in skin from baseline to 4 weeks | 0 and 4 weeks

SECONDARY OUTCOMES:
change in lipid profile (TG, Chol, LDL, HDL, ox LDL, glycated LDL, fattyacids)from baseline to 4 weeks | 0 and 4 weeks
change in HbA1c from baseline to 4 weeks | 0 and 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Susanne G Bugel, Principal Investigator — Department of Human Nutrition, University of Copenhagen
Locations (1):
- Department of Human Nutrition, University of Copenhagen, Frederiksberg, Denmark